CLINICAL TRIAL: NCT02648867
Title: Evaluation of Continuous Maternal Feedback to Shorten Second Stage Labor
Brief Title: Evaluation of Maternal Feedback to Shorten Pushing Efforts During Labor
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device was unacceptable to patients and did not provide expected outputs
Sponsor: Clinical Innovations, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CI-002-PC
Record Dates: First submitted 2016-01-03; First posted 2016-01-07 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Prolonged Second Stage of Labor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients receiving PushCoach feedback (Experimental): Patients will receive continuous maternal feedback from the PushCoach device, which includes both audio and visual feedback of fetal head movement during the second stage of labor
  Interventions: Device: Continuous Maternal Feedback
- Patients blinded to PushCoach feedback (Active Comparator): Patients will not receive continuous maternal feedback from the PushCoach device (it will be in place and collect data), but will receive normal feedback from the clinician during the second stage of labor.
  Interventions: Device: Continuous Maternal Feedback

INTERVENTIONS:
Device: Continuous Maternal Feedback — The PushCoach device consists of a modification of the standard fetal scalp electrode and a separate apparatus designed to detect movement of the fetal head by detecting movement of an FSE. The PushCoach will be attached to the patient by an adhesive pad over the sacrum and extend between the patient's legs approximately 2-3 inches from the vaginal introitus. It assesses the movement of the FSE attached to the fetal scalp during pushing. The amount of fetal movement will be measured and recorded. The PushCoach device is connected to a laptop computer which will provide optical and auditory feedback to the patient about descent of the fetal head with maternal expulsive efforts.
  Other Names: PushCoach

SUMMARY:
This study will assess the ability for continuous electronic feedback to reduce the length of second stage labor and improve maternal and fetal outcomes.

DETAILED DESCRIPTION:
The length of the second stage (pushing stage) of labor is highly correlated with the incidence of adverse outcomes for mother and neonate. More than 80% of laboring women in the US have epidurals for labor pain management. The length of second stage labor is increased in women receiving regional anesthesia for pain management during labor and delivery compared to women without anesthesia. This increased length of labor is largely due to lack of maternal sensation resulting in decreased physiologic feedback on the efficacy of maternal expulsive (pushing) efforts. Continuous maternal feedback regarding fetal decent during labor may result in more effective maternal expulsive efforts reducing the length of second stage and improving maternal and neonatal outcomes. This study will assess the ability for continuous electronic feedback to reduce the length of second stage labor and improve maternal and fetal outcomes.

The study device consists of a modification of the standard fetal scalp electrode and a separate apparatus designed to detect movement of the fetal head by detecting movement of the FSE. As the patient pushes, the amount of fetal movement will be measured and recorded. The movement will be recorded by a laptop computer which will provide optical and auditory feedback to the patient about descent of the fetal head with maternal expulsive efforts.

ELIGIBILITY:
Inclusion Criteria:

1. Laboring nulliparous women who are > 36 0/7 weeks estimated gestational age undergoing epidural or combined spinal epidural (CSE) placement for labor pain management.

Exclusion Criteria:

1. Women with multiple gestations.
2. Women with contraindications to pushing during second stage labor.
3. Women with contraindications to Fetal Spiral Electrode (FSE) placement including women with a face or compound presentation, known HIV, Hepatitis B or Active Herpes.
4. Women who do not plan to initiate pushing immediately (those who plan to "rest and descend" prior to initiation of pushing).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Length of second stage labor in patients using the PushCoach device compared to patients blinded to the PushCoach device output | Second stage of labor begins once the patient's cervix is completely dilated and ends once the baby is delivered. This time will be compared between patients.
  The primary objective of this study is to measure the ability of immediate, quantitatively precise, visual, and auditory and haptic maternal feedback on fetal descent to reduce the overall length of second stage labor compared to women receiving standard verbal and manual feedback during second stage labor and reduce the incidence of pushing for longer than 60 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Esplin, M.D., Principal Investigator — Intermountain Health Care, Inc.; Erin Clark, M.D., Principal Investigator — University of Utah Hospital; George Saade, M.D., Principal Investigator — University of Texas
Locations (3):
- United States (3):
  - University of Texas Medical Branch, Galveston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Intermountain Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McRae-Bergeron CE, Andrews CM, Lupe PJ. The effect of epidural analgesia on the second stage of labor. AANA J. 1998 Apr;66(2):177-82. PMID 9801480
- [Background] Johnson S, Rosenfeld JA. The effect of epidural anesthesia on the length of labor. J Fam Pract. 1995 Mar;40(3):244-7. PMID 7876781
- [Background] Rouse DJ, Weiner SJ, Bloom SL, Varner MW, Spong CY, Ramin SM, Caritis SN, Peaceman AM, Sorokin Y, Sciscione A, Carpenter MW, Mercer BM, Thorp JM Jr, Malone FD, Harper M, Iams JD, Anderson GD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Second-stage labor duration in nulliparous women: relationship to maternal and perinatal outcomes. Am J Obstet Gynecol. 2009 Oct;201(4):357.e1-7. doi: 10.1016/j.ajog.2009.08.003. PMID 19788967